CLINICAL TRIAL: NCT01490411
Title: A Randomized, Double Blind, Placebo-Controlled, Parallel Group Study to Investigate the Relative Efficacy and Safety of Immunotherapy With rBet v1-FV Compared to Placebo in Birch Pollen-Allergic Patients With IgE-Mediated Seasonal Allergic Rhinoconjunctivitis
Brief Title: Dose Range Finding Study With rBet v1-FV - in Adult Patients With Birch Pollen-Allergic Seasonal Rhinoconjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL0903rB; P2IX09001 (Other: CETERO RESEARCH)
Record Dates: First submitted 2011-11-18; First posted 2011-12-13 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: Specific immunotherapy; SIT; SCIT; recombinant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Placebo was given the same way as a subcutaneous (just under the skin) injection. Patients received at least 10 injections of Placebo or rBet v1-FV.
  Interventions: Drug: Placebo
- 20 µg rBet v1-FV Immunotherapy (Experimental): The drug tested in this study (rBet v1-FV) was given as a subcutaneous (just under the skin) injection. Patients received at least 10 injections of Placebo or rBet v1-FV, administered in increasing doses weekly for 10 weeks, up to one of the maximum concentrations.
  Interventions: Biological: rBet v1-FV
- 80 µg rBet v1-FV Immunotherapy (Experimental): The drug tested in this study (rBet v1-FV) was given as a subcutaneous (just under the skin) injection. Patients received at least 10 injections of Placebo or rBet v1-FV, administered in increasing doses weekly for 10 weeks, up to one of the maximum concentrations.
  Interventions: Biological: rBet v1-FV
- 160 µg rBet v1-FV Immunotherapy (Experimental): The drug tested in this study (rBet v1-FV) was given as a subcutaneous (just under the skin) injection. Patients received at least 10 injections of Placebo or rBet v1-FV, administered in increasing doses weekly for 10 weeks, up to one of the maximum concentrations.
  Interventions: Biological: rBet v1-FV
- 320 µg rBet v1-FV Immunotherapy (Experimental): The drug tested in this study (rBet v1-FV) was given as a subcutaneous (just under the skin) injection. Patients received at least 10 injections of Placebo or rBet v1-FV, administered in increasing doses weekly for 10 weeks, up to one of the maximum concentrations.
  Interventions: Biological: rBet v1-FV

INTERVENTIONS:
Drug: Placebo — The drug tested in this study (rBet v1-FV) was given as a subcutaneous (just under the skin) injection. Patients received at least 10 injections of Placebo or rBet v1-FV, administered in increasing doses weekly for 10 weeks, up to one of the maximum concentrations.
  Other Names: Comparator
  Arms: Placebo
Biological: rBet v1-FV — The drug tested in this study (rBet v1-FV) was given as a subcutaneous (just under the skin) injection. Patients received at least 10 injections of Placebo or rBet v1-FV, administered in increasing doses weekly for 10 weeks, up to one of the maximum concentrations.
  Other Names: Specific Immunotherapy
  Arms: 20 µg rBet v1-FV Immunotherapy
Biological: rBet v1-FV — The drug tested in this study (rBet v1-FV) was given as a subcutaneous (just under the skin) injection. Patients received at least 10 injections of Placebo or rBet v1-FV, administered in increasing doses weekly for 10 weeks, up to one of the maximum concentrations.
  Other Names: Spicific Immunotherapy
  Arms: 80 µg rBet v1-FV Immunotherapy
Biological: rBet v1-FV — The drug tested in this study (rBet v1-FV) was given as a subcutaneous (just under the skin) injection. Patients received at least 10 injections of Placebo or rBet v1-FV, administered in increasing doses weekly for 10 weeks, up to one of the maximum concentrations.
  Other Names: Specific Immunotherapy
  Arms: 160 µg rBet v1-FV Immunotherapy
Biological: rBet v1-FV — The drug tested in this study (rBet v1-FV) was given as a subcutaneous (just under the skin) injection. Patients received at least 10 injections of Placebo or rBet v1-FV, administered in increasing doses weekly for 10 weeks, up to one of the maximum concentrations.
  Other Names: Spicific Immunotherapy
  Arms: 320 µg rBet v1-FV Immunotherapy

SUMMARY:
The purpose of this study is to find out if rBet v1-FV works to relieve Seasonal Allergic Rhinitis symptoms compared to Placebo (an inactive substance that looks like rBet v1-FV and also contains Aluminum Hydroxide but does not contain the experimental drug). rBet v1-FV is a vaccine that works by exposing your immune system to something that resembles birch. This vaccine may help to lessen your allergy symptoms during the natural birch season.

DETAILED DESCRIPTION:
Type I allergy is an immune-disorder which stems from the formation of IgE antibodies against proteins and glycoproteins from plants, insects, animals and fungi, most of which are normally considered harmless. The cross-linking of specific IgE antibodies on effector cells by allergens activates an immunological cascade leading to the symptoms of Type I allergy including rhinitis, conjunctivitis, asthma, and anaphylactic shock. Allergic Rhinitis is the most common chronic atopic disease and is associated with considerable cost and co-morbidity. Seasonal allergic rhinitis (SAR), triggered by pollen from trees, grasses and weeds, is characterized by sneezing, nasal congestion, nasal itching, rhinorrhea, and pruritic, watery, red eyes.

Recombinant preparations offer various advantages over those based on natural allergen extracts. Recombinant proteins can be produced in highly purified forms of pharmaceutical quality; proteins are molecularly defined thus ensuring product consistency and minimising problems related to allergen extract standardisation; preparations only include those proteins that are considered relevant for specific immunotherapy; the risk of contamination with other allergenic material is excluded; the whole production process can be designed to exclude any risk factors for the introduction of infectious agents; the relative dosages of individual components of a final preparation can be optimised to favour better clinical efficacy. Allergy vaccination (AV) mediates the immune response to allergen exposure by altering the TH2 response in favour of a TH1 T-cell response, increasing IgG production and decreasing the production of inflammatory cytokines. rBet v1-FV is an AV designed to enhance beneficial immune responses. The investigational product has demonstrated efficacy and good tolerability in one previous pivotal Phase III and two previous Phase II studies.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following to be eligible for enrollment:

* Is a male or female, aged 18 to 65 years, inclusive.
* Has a clinical history of allergic rhinitis to birch pollen at least during each of the last 2 years.
* Has a birch pollen specific IgE result (EAST) greater than 0.75 kU/L on blood sample drawn at Visit 1.
* Has a positive skin prick test to birch allergen(s) at Visit 1, with a wheal diameter of at least 4 mm.
* Has minimum qualifying symptom scores at Visit 2.
* Patients with sensitization to cat epithelia, dog epithelia, Dermatophagoides farinae or Dermatophagoides pteronyssinus as per the skin prick test and/or EAST, may be included if sensitization is not clinically relevant.
* Meets the concomitant medication restrictions described in the protocol.
* Is normally active and otherwise judged to be in good health on the basis of medical history, physical examination and routine laboratory tests.
* Is willing and able to give signed informed consent, and must have provided this consent.
* Is willing and able to attend required study visits.

Exclusion Criteria:

A patient will not be included in this study if any of the following criteria apply:

For female subjects:

* Female subjects with childbearing potential (i.e., females are not chemically or surgically sterilised or females who are not post-menopausal) with a positive pregnancy test at Visit 1.
* Female subjects with a negative pregnancy test at enrolment and not willing to use a reliable and highly effective method of birth control with a low failure rate (i.e. less than 1% per year) when used consistently and correctly during the trial, as judged by the investigator.
* Pregnancy and lactation.
* Female subjects seeking to become pregnant.

General criteria:

* Individuals weighing less than 40 Kg.
* Not able to understand and comply with the requirements of the trial, as judged by the investigator.
* Concurrent participation in any other clinical trial or participation in any other clinical trial during the previous 30 days.
* Treatment with beta-blockers (locally and systemically).
* Contraindication for adrenalin (e.g. acute or chronic symptomatic coronary heart disease, severe hypertension).

Immunotherapy criteria:

* Previous specific immunotherapy with birch or other early blossoming trees (e.g. Alder, Hazel) in any formulation within the past 5 years.
* Any current immunotherapy.
* Any previous specific immunotherapy with unknown or mixed allergens.

Other allergies:

- Clinically relevant perennial allergies.

Diseases and health status:

* Clinically relevant rhinoconjunctival or respiratory symptoms related to other reasons.
* Has diagnosed asthma.
* Has PEF or FEV1 < 80% of predicted normal
* Any acute or chronic disease that, in the opinion of the investigator, would affect the study objectives or subject safety (e.g., Diabetes mellitus type I, malignant neoplasia, chronic renal failure, inflammatory diseases of liver or kidneys, emphysema, bronchiectasis).
* Autoimmune diseases, immune-defects including immune-suppression, immune-complex-induced immunopathies (e.g. HIV, post-transplant patients, lupus erythematodes [SLE], Grave's disease, Hashimoto's thyroiditis) at time of screening.
* Has a history of other clinically significant diseases which might impact efficacy analysis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Relative efficacy of four different doses compared to placebo. | 6 hours
  To assess the relative efficacy of four different dose regimes of rBet v1-FV compared to Placebo based on post-treatment intracutaneous testing results. The post-treatment wheal size (length in mm) after intracutaneous injection of a birch pollen solution was determined.

SECONDARY OUTCOMES:
Relative efficacy of four different dose regimes of rBet v1-FV compared to Placebo and to each other in the reduction of symptoms of allergic rhinitis in the Environmental Exposure Chamber (EEC). | 1, 2, 3, 4, 5, 6, 7 and 8.0 hour(s) in the EEC
  To assess the relative efficacy of four different dose regimes of rBet v1-FV compared to Placebo and to each other in the reduction of symptoms of allergic rhinitis in the Environmental Exposure Chamber (EEC), based on the change from baseline in area under the curve (AUC) for Total Symptom Score (TSS), Total Nasal Symptom Score (TNSS), Total Non-Nasal Symptom Score (TNNSS) and Total Ocular Symptom Score (TOSS).
Relative safety and tolerability of four different dose regimes of rBet v1-FV compared to Placebo | 3-12 month
  Recording of all adverse events, the vital signs and clinical laboratory tests.

CONTACTS AND LOCATIONS:
Overall Officials: Deepen Patel, MD, CCFP, Principal Investigator
Locations (1):
- Allergopharma GmbH & Co. KG, Hamburg, Reinbek, Germany

REFERENCES:
- [Result] Meyer W, Narkus A, Salapatek AM, Hafner D. Double-blind, placebo-controlled, dose-ranging study of new recombinant hypoallergenic Bet v 1 in an environmental exposure chamber. Allergy. 2013 Jun;68(6):724-31. doi: 10.1111/all.12148. Epub 2013 Apr 27. PMID 23621350